CLINICAL TRIAL: NCT04233983
Title: Surgery Before Embryo Transfer in Endometrioma Related Reduction in Ovarian Reserve
Brief Title: Surgery Before Embryo Transfer in ERROR (Endometrioma Related Reduction in Ovarian Reserve)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, GÜRKAN UNCU,PROF. MD, Prof. Dr., Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-19/12
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Endometriosis Related Infertility
Keywords: Endometriosis; Laparoscopy; Infertility; Ovarian Reserve; Endometrioma
MeSH Terms: conditions — Endometriosis; Infertility

STUDY DESIGN:
Intervention Model Description: Prospective Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): The study group consists of ERROR(endometrioma related reduction in ovarian reserve) patients who will undergo laparoscopic endometriosis surgery after ICSI procedure with freezing all embryos. The patients will wait about 6 months for spontaneous conception, if there is no pregnancy during this period, frozen embryo transfer will be performed.
  Interventions: Procedure: Laparoscopic Endometriosis Surgery
- Control Group (No Intervention): The control group consists of ERROR(endometrioma related reduction in ovarian reserve) patients who will be performed IVF&ICSI procedure with fresh embryo transfer without surgery. If there is no pregnancy, patients will be operated then.

INTERVENTIONS:
Procedure: Laparoscopic Endometriosis Surgery — Patient with ERROR(endometrioma related reduction in ovarian reserve), and endometrioma larger than 3 cm diameter will be operated after IVF&ICSI procedure. Operation will be done by senior surgeons of our department. Laparoscopic endometrioma operation procedure consists of excision of endometrioma cyst with its capsule from ovary without using any electric modality to prevent ovarian damage.
  Arms: Study Group

SUMMARY:
This prospective study evaluates the pregnancy results after laparoscopic endometriosis operation in infertile patients with ERROR (endometrioma related reduction in ovarian reserve)

DETAILED DESCRIPTION:
This study consists of two groups. Patients will be randomly enrolled into the groups by ART (assisted reproductive technology) centre nursery. All patients will sign a consent form about procedure.

Patients diagnosed with endometrioma (larger than 3 cm diameter) and ERROR (endometrioma related reduction in ovarian reserve - Antimullerian Hormon < 1.2 ng/ml, Antral follicle count < 7 , Day3 Follicle Stimulating Hormone > 10 IU/dl, Low response to ovarian hyper stimulation < 3 oocytes) will be enrolled in study. Patients with age >40, with male factor, with undefined adnexal mass, malignity suspicion will be excluded from study.

The study group consists of patients who will undergo laparoscopic endometriosis surgery after ICSI procedure with freezing all embryos. The patients will wait about 6 months for spontaneous conception, if there is no pregnancy during this period, frozen embryo transfer will be performed. The control group consists of patients who will be performed IVF&ICSI procedure with fresh embryo transfer without surgery. If there is no pregnancy, patients will be operated then.

As the primary; result positive b-hCG rates will be compared between groups.

In conclusion we will find out whether laparoscopic endometriosis operation improves or worsens the pregnancy results in patients with ERROR.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Endometrioma at least in one ovary, larger than 3 cm diameter
* Endometriosis Related Reduction in Ovarian Reserve (ERROR)
* Presence of endometriosis related infertility

Exclusion Criteria:

* Presence of chronic systemic disease
* Presence of male factor infertility
* Suspicion of ovarian malignancy or undefined ovarian mass

Ages: 23 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Positive b-hCG Rate | 6 months
  Postoperative 6. months positive b-hCG rates will be compared with control group.

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Uncu, Prof., Study Director — Bursa Uludag University School of Medicine ART Center
Locations (1):
- Uludag University ART Center, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muzii L, Di Tucci C, Di Feliciantonio M, Marchetti C, Perniola G, Panici PB. The effect of surgery for endometrioma on ovarian reserve evaluated by antral follicle count: a systematic review and meta-analysis. Hum Reprod. 2014 Oct 10;29(10):2190-8. doi: 10.1093/humrep/deu199. Epub 2014 Aug 1. PMID 25085800
- [Result] Kasapoglu I, Ata B, Uyaniklar O, Seyhan A, Orhan A, Yildiz Oguz S, Uncu G. Endometrioma-related reduction in ovarian reserve (ERROR): a prospective longitudinal study. Fertil Steril. 2018 Jul 1;110(1):122-127. doi: 10.1016/j.fertnstert.2018.03.015. Epub 2018 Jun 20. PMID 29935810